CLINICAL TRIAL: NCT00713024
Title: Patterns of Cerebral Activation to Innocuous and Noxious Heat Stimulations in Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sung-Tsang Hsieh, Department of Neurology, National Taiwan University Hospital
Other Study IDs: 200712022R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Neuropathic Pain
Keywords: Pain; Functional neuroimaging; Neuropathy; Thermal sensation
MeSH Terms: conditions — Neuralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Healthy control subjects
- 2: Patients having neuropathic pain

SUMMARY:
Patients with neuropathic pain exhibit hyperalgesia and allodynia. Although both peripheral and central determinants are recognized for the pathophysiological basis of neuropathic pain following peripheral injury, the modulating effect on pain processing in brain by peripheral mechanisms remains elusive. Here, we will systematically compare the sensory symptoms and brain activation to innocuous and noxious thermal stimulation applied to the distal leg, foot dorsum or forearm between patients with peripheral neuropathy and healthy controls. Functional magnetic resonance imaging will be used to define brain activation to somatic stimulation with noxious and innocuous stimuli. The blood-oxygenation-level-dependent signals will be correlated with visual analogue scale scores and sensory and affective components obtained from the Short-Form McGill Pain Questionnaire. Brain activation during thermal stimulation in patients with neuropathic pain will be clarified, and we will also analyze the potential relationships between the topography, quality and intensity of the different painful symptoms (i.e. spontaneous ongoing pain, paroxysmal pain, allodynia, hyperalgesia) and the magnitude and pattern of brain activation during thermal stimulation. This will add in our understanding in the pathophysiology of brain modulation in pain and provide clinically useful message toward the potential therapeutics in the management of neuropathic pain.

DETAILED DESCRIPTION:
Many patients with neuropathic pain exhibit hyperalgesia and allodynia. In various pain syndromes, neuropathic pain is among the most difficult to treat. Previous studies show that the development of secondary hyperalgesia results from abnormal processing of nociceptor input after injuries of the peripheral nervous system. However, the modulating effect on pain processing in brain by peripheral mechanisms remains elusive, and only few studies investigate the issue.

Evidences suggest that lesions of the spinothalamocortical pathway may be necessary for developing the central pain, indicating indirect changes in excitability due to alterations of pain modulatory systems. Previous anatomical, physiological, and lesion studies have revealed an extensive cortical network associated with sensory, cognitive, and affective aspects of pain, including primary somatosensory cortex, secondary somatosensory cortex, insular cortex, and anterior cingulate cortex. Moreover, a recent study reported that neuropathic pain might influence brain organization. Therefore, it would be intriguing to know whether and how the brain processes pain in patients with neuropathic pain.

We hypothesize that neuropathic pain elicited by the peripheral neuropathy results in hyperexcitability of the pain matrix (i.e. central sensitization) due to alterations of pain modulatory systems. Patients with peripheral neuropathy and healthy volunteers will be recruited in this study. Peripheral neuropathy is defined according to the neuropathic symptoms and signs. For healthy volunteers, clinical history will be evaluated by questionnaires and neurological examinations to exclude any neuropsychiatric disorder or pain condition.

To assess the severity of different neuropathic symptoms,patients with neuropathic pain will fill out the Neuropathic Pain Symptom Inventory (NPSI). Each subject will receive detailed sensory examination to evaluate the integrity of small-diameter and large-diameter sensory fibers. To measure thresholds of thermal and vibratory sensations, we will perform quantitative sensory testing (QST) by the method of level using a Thermal Sensory Analyser and Vibratory Sensory Analyser (Medoc Advanced Medical System, Minneapolis, MN, USA) following an established protocol. Thermal thresholds will be recorded on the toe, and vibratory thresholds recorded on the lateral malleolus. These values will be compared with normative values for the age, which had been documented previously.

Functional magnetic resonance imaging (fMRI) will be performed on a 3-T MR machine (Trio; Siemens, Erlangen, Germany). A high resolution T1 weighted scan of the entire brain in trans-axial orientation will be obtained to provide anatomical information for the superimposed functional activation maps. Echo Planar Imaging will be used for the acquisition of the functional data.

We will use a CHEP stimulator (Medoc Ltd, Ramat Yishai, Israel) to deliver thermal stimulation. The 27 mm diameter thermode is comprised of a heating thermofoil (Minco Products, Inc., Minneapolis, MN) that is covered with a thermoconductive plastic. The stimulus temperatures given throughout this report will be referred to the temperature of the thermofoil. Cooling will begin immediately following attainment of the pre-fixed target temperature. Individual heat pain threshold (HPT) will be measured before fMRI scans. Noxious heat and innocuous heat will be applied within the distal leg, foot dorsum or forearm. The thermode will be remained at the same site during each block of functional MRI scans. Several pretests will be applied before CHEP recording to eliminate expectation effects. To avoid sensitization and desensitization, low intensity stimuli will precede high intensity stimuli at each block.

Each imaging session will be consisted of one high-resolution anatomical scan and three functional scanning runs, with 5-min intersession interval. During the scanning, five thermal stimuli will be applied by CHEP stimulator to the right dorsal foot. To avoid sensitization, habituation and tissue damage, the stimulation temperature will be applied in a random fashion, and the stimulation site will be changed slightly after each stimulus. After 12-s stimulation, the temperature will be cooling, with a subsequent 36-s interstimulus interval. After each fMRI session, subjects will be asked to rate the intensity and unpleasantness of received pain stimulus. The average rating values will be indicated after the scan on a computer driven visual analogue scale (VAS) ranging from 0 to 10 (0, no sensation; 1, slight intense; 2, innocuous warmth; 3, innocuous heat; 4, slight pain; 5, mild pain; 7, moderate-strong pain; 9, severe pain; 10, unbearable pain), and the intensity and unpleasantness of received pain will be assessed using the Short-Form McGill Pain Questionnaire (SFMPQ).

All data will be processed using the Statistical Parametric Mapping software (SPM2, Wellcome Department of Cognitive Neurology, London UK). fMRI data series will be realigned and resliced with sinc interpolation to correct for motion artifacts. Scans with sudden head movements of more than 2 mm will be omitted. To enable intersubject analysis, the functional data will be coregistered to the anatomical scan and transformed into a reference space according to the MNI template of SPM2 by normalization using sinc interpolation. This template has been determined from 305 MRI scans of healthy subjects at the Montreal Neurological Insitute. The resampled voxel volume of the normalized images is 2 x 2 x 2 mm. Subsequently, data will be smoothed with an isotropic Gaussian kernel of 8 mm full-width at half maximum to reduce high frequency noise and to account for anatomical variances. Condition-specific effects will be estimated with the general linear model using a boxcar approach convolved with the hemodynamic response function. High pass filtering will remove low frequency noise and low pass filtering will account for serial autocorrelations of the data.

We will analyze the data on an individual (subject per subject) basis and across subjects (group analysis) using a cross-subjects variance (random effect analysis). We will compute different contrasts between cerebral responses during innocuous and noxious heat stimulation. Data from each stimulation will be pooled for group statistical comparisons. A group activation map will be constructed by performing a conjunction analysis to measure the spatial overlap of activation across subjects. A single design matrix, including 3 sessions of all subjects, will be generated due to the limited number of experiments representing a fixed-effects model analysis. Statistical parametric maps will be generated as t-contrasts and corrected for multiple comparisons according to the random field theory with P < 0.05. The threshold for the Z maps is 3.09 (P < 0.001) for individual subject analysis. Significant clusters have to show a minimum extension volume of 10 voxels. For group analysis, parametric maps will be constructed using the same contrast and spatial extent but we will use a corrected threshold of P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients having neuropathic pain
* healthy control subjects

Exclusion Criteria:

* subjects with pacemaker implantation
* patients with neuropsychiatric disorder except neuropathic pain
* subjects with agoraphobia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit healthy control subjects and patients having neuropathic pain in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, MD, PhD, Study Director — Department of Neurology, National Taiwan University Hospital
Locations (1):
- Department of Neurology, National Taiwan University Hospital, Taipei, Taiwan